CLINICAL TRIAL: NCT06209346
Title: Multimodal Physiotherapy Based on Tele-rehabilitation in Chronic Pelvic Pain Associated With Endometriosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Maria Torres Lacomba, Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEID/2023/6/106
Record Dates: First submitted 2023-12-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-07

CONDITIONS: Endometriosis; Chronic Pelvic Pain Syndrome
Keywords: endometriosis; chronic pelvic pain; physical therapy; pain education
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TeleRehab Group (Experimental): The duration of treatment for the TeleRehab Group will be 8 weeks and will consist of a total of 20 sessions, with between 2 and 3 sessions per week depending on the week they are in.
  Weeks 2, 4, 6 and 8 will have 2 sessions per week and weeks 1, 3, 5 and 7 will have 3 sessions per week.
  These sessions will consist of videos that will make up the educational material, videos that will guide the TE program and respiratory control practices. All the sessions mentioned above will be in online format, through the TRAK platform.
  Interventions: Other: TeleRehab Group
- Advices Group (Active Comparator): They will receive informative material in weeks 1, 3, 5 and 7 about their pathology and with recommendations for them to achieve healthy lifestyle habits that do not further damage their disease. o Participants in the Advices Group will have the same follow-up assessments as the TeleRehab Group and will receive informative material. They will not have access to the audiovisual material generated for the TeleRehabGroup.
  Interventions: Other: Advices Group

INTERVENTIONS:
Other: TeleRehab Group — The duration of treatment for the Experimental Group will be 8 weeks and will consist of a total of 20 sessions, with between 2 and 3 sessions per week depending on the week they are in.
  Weeks 2, 4, 6 and 8 will have 2 sessions per week and weeks 1, 3, 5 and 7 will have 3 sessions per week.
  These sessions will consist of videos that will make up the educational material, videos that will guide the ET program and respiratory control practices.All the sessions mentioned above will be in online format, through the TRAK platform.
  Other Names: TrhbG
  Arms: TeleRehab Group
Other: Advices Group — They will receive informative material in weeks 1, 3, 5 and 7 about their pathology and with recommendations for them to achieve healthy lifestyle habits that do not further damage their disease. Participants in the Control Group will have the same follow-up evaluations as the Experimental Group and will receive informative material. They will not have access to the audiovisual material generated for the Experimental Group.
  Other Names: AG
  Arms: Advices Group

SUMMARY:
* Objective: To determine if the tele-rehabilitation program for chronic pelvic pain associated with endometriosis composed of pain education, therapeutic exercise and respiratory control decreases pain according to the Visual Numerical Scale (EVN), catastrophizing with the Pain Catastrophizing Scale (PCS), kinesiophobia with the Tampa Scale of Kinesiophobia (TSK), improves sexual function according to the Female Sexual Function Index (FSFI) and QoL compared to the Control Group with the Health Status Questionnaire (SF-12).
* Follow-up: four evaluated questionnaires: preintervention; postintervention, 3 months postintervention, 6 months postintervention
* Participants: 66 women diagnosed with endometriosis with chronic pelvic pain in different Spanish endometriosis associations.
* Randomization: women will be randomly assigned to two groups using the EpiData 3.1 software
* Interventions: Experimental Group: therapeutic exercise + conscious breathing (16 sessions) and pain education (4 sessions) through the TRAK platform.

Control Group: They will receive informative material in weeks 1, 3, 5 and 7 about their pathology and with recommendations for them to achieve healthy lifestyle habits that do not further damage their disease.

ELIGIBILITY:
Inclusion Criteria:

* Women with a medical diagnosis of endometriosis.
* Age equal to or older than 18 years and up to 55 years.
* Who are or have received medical and/or surgical treatment and with controlled disease.
* Persistent pelvic pain for at least 3 months.
* Pain greater than 4 on the EVN.
* No cognitive limitation to understand the information sheet, instructions and freely sign the informed consent
* Have any electronic device available (tablet, computer, cell phone).
* Have a current email address.
* Have a valid e-mail address.

Exclusion Criteria:

* Peri- and postmenopausal women.
* Women pregnant or desiring gestation during the study.
* Women with a history of gynecologic cancer and/or undergoing any systemic and/or localized oncologic treatment in the pelviperineal region
* Women with a diagnosis of chronic fatigue or fibromyalgia▪.
* Women concomitantly participating in another intervention study.
* Women undergoing surgery during the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 66 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-01-17 (Estimated); Study Completion 2027-01-17 (Estimated)

PRIMARY OUTCOMES:
Health Status Questionnaire (SF-12) | Pre-intervention (baseline); Post-intervention (two month from baseline); and 3 and 5 months post-intervention. A score of 0 means poorer health and a score of 100 means better health.
  Change from baseline in quality of life at two month (post-intervention); and 3 and 5 months post-intervention
Visual Numeric Scale (VNS) | Pre-intervention (baseline); Post-intervention (two month from baseline); and 3 and 5 months post-intervention. A score of 0 means no pain, 1 to 3 means mild pain, 4 to 6 means moderate pain and 7 to 10 means severe pain.
  Change from baseline in pain at two month (post-intervention); and 3 and 5 months post-intervention
Endometriosis Health Profile (EHP-30) | Pre-intervention (baseline); Post-intervention (two month from baseline); and 3 and 5 months post-intervention. A score of 0 indicates the best health status to the worst health status of 100.
  Change from baseline in endometriosis affectation at two month (post-intervention); and 3 and 5 months post-intervention
Index of Sexual Function (IFSF) | Pre-intervention (baseline); Post-intervention (two month from baseline); and 3 and 5 months post-intervention. The final score (total score: minimum 2 and maximum 36). The higher the better sexual function, the lower the worse sexual function.
  Change from baseline in sexual function at two month (post-intervention); and 3 and 5 months post-intervention
Tampa Scale of Kinesiophobia (TSK) | Pre-intervention (baseline); Post-intervention (two month from baseline); and 3 and 5 months post-intervention. The lowest possible score, 11, no kinesiophobia. The highest possible score, 44, denotes a severe kinesophobia
  Change from baseline in kinesiophobia at two month (post-intervention); and 3 and 5 months post-intervention
Pain Catastrophizing Scale (PCS) | Pre-intervention (baseline); Post-intervention (two month from baseline); and 3 and 5 months post-intervention. The overall score has a range of 0-52. Higher scores indicate a greater degree of pain catastrophizing.
  Change from baseline in catastrophixing at two month (post-intervention); and 3 and 5 months post-intervention

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Pre-intervention (baseline); Post-intervention (two month from baseline); and 3 and 5 months post-intervention. The overall score ranges from 0 to 21 points. Normal range (0-7), Possible A/D (8-10) and Case A/D
  Change from baseline in anxiety and depression at two month (post-intervention); and 3 and 5 months post-intervention
International Physical Activity Questionnaire (IPAQ) | Pre-intervention (baseline); Post-intervention (two month from baseline); and 3 and 5 months post-intervention. Low: low physical activity Medium: 3+days of vigorous physical activity.High:performs vigorous physical activity reaching a high energy
  Change from baseline in physical activity at two month (post-intervention); and 3 and 5 months post-intervention
Pittsburg Sleep Quality Index (PSQI) | Pre-intervention (baseline); Post-intervention (two month from baseline); and 3 and 5 months post-intervention. The overall score ranges from 0 (no difficulty) to 21 (difficulties in all areas).
  Change from baseline in sleep quality at two month (post-intervention); and 3 and 5 months post-intervention
Perceived Stress Scale (PSS) | Pre-intervention (baseline); Post-intervention (two month from baseline); and 3 and 5 months post-intervention. The score ranges from 0 to 56 and indicates that a higher score corresponds to a higher level of perceived stress.
  Change from baseline in stress at two month (post-intervention); and 3 and 5 months post-intervention
Patient's adherence will be evaluated | Pre-intervention (baseline); Post-intervention (two month from baseline); and 3 and 5 months post-intervention
  Adherence (via TRAK Platform with email and chat)
Patient global impression of change (PGI-I) | Pre-intervention (baseline); Post-intervention (two month from baseline). The score ranges from 1 to 7 and indicates that a higher score corresponds to worsening with treatment and a lower score to improvement with treatment.
  Patient global impression of change (PGI-I)

OTHER OUTCOMES:
Body mass index (BMI) | Pre-intervention (baseline); Post-intervention (two month from baseline); and 3 and 5 months post-intervention.
  BMI can give a general idea of whether a person is at a healthy weight and It is important to know how this relates to endometriosis and pain
Employment status | Pre-intervention (baseline)
  It is important to know the patient's current work status for her medical history and how this relates to endometriosis and pain
Education level | Pre-intervention (baseline)
  It is important to know the patient's educational level for her medical history and how this relates to endometriosis and pain.
Ethnicity | Pre-intervention (baseline)
  It is important to know the patient's ethnicity for her medical history and how this relates to endometriosis and pain.
Maritial status | Pre-intervention (baseline)
  It is important to know the patient's marital status for her medical history and how this relates to endometriosis and pain.
Number of children | Pre-intervention (baseline)
  It is important to know if and how many children the patient has for her medical history and how this relates to endometriosis and pain.
Age | Pre-intervention (baseline); Post-intervention (two month from baseline); and 3 and 5 months post-intervention.
  It is important to know the patient's age for her medical history and how this relates to endometriosis and pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Physiotherapy in women´s health research group. University of Alcalà, Alcalà de Henares, Madrid, Spain